CLINICAL TRIAL: NCT02886182
Title: Immune Function Status and the Prevalence of Hepatitis in Postpartum Pregnant Women With Chronic Hepatitis B Virus Infection
Brief Title: Immune Function Status and the Prevalence of Hepatitis in Postpartum Pregnant Women With CHB Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY010
Record Dates: First submitted 2016-08-19; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; pregnancy; Cellular immune response; Clinical implications
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Keeping the serum samples frozen at - 80℃low temperature refrigerator preservation to detect cytokine by high flux liquid chip technology (Luminex)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group A: pregnants who were positivity for serum HBsAg for more than 6 months and HBeAg , HBV DNA >106IU/mL, alanine aminotransferase (ALT) below 35 IU/mL (ULN=40IU/mL) and no received nucleoside analogue antiviral therapy were enrolled into group A
- group B: the CHB infection pregnants with undetectable HBVDNA were enrolled into group B(control group)

SUMMARY:
To date, several studies have manifested that high levels of adrenal corticosteroids and oestrogen hormones during pregnancy can lead to increased HBV viraemia. These hormonal and immune function status changes can result in minimal fluctuations in liver function tests. Serum alanine aminotransferase (ALT) tends to increase in late pregnancy and the postpartum period. Peripartum hepatitis flares leading to hepatic decompensation have been reported.Therefore, the investigators aim to detect and observe the immune function status and incidence of hepatitis in pregnant women with chronic hepatitis B virus infection in late pregnancy and the postpartum period.To provide a clinical evidence for the administration of chronic hepatitis B virus infection pregnant women.

DETAILED DESCRIPTION:
In this trial, pregnants who were positivity for serum HBsAg for more than 6 months and HBeAg , HBV DNA >106IU/mL, alanine aminotransferase (ALT) below 35 IU/mL (ULN=40IU/mL) and no received nucleoside analogue antiviral therapy were enrolled into group A, In addition ,the CHB infection pregnants with undetectable HBVDNA were enrolled into group B(control group).In which, all pregnants were chronic HBV infection without compensated cirrhosis,hepatic adipose infiltration,ICP, hypertension ,heart disease, postpartum hemorrhage. None of the mothers were co-infected with hepatitis A,C,D,E,or HIV;syphilis, Epstein-Barr virus.Serum HBV DNA load(Roche, Pleasanton, CA, USA), HBsAg/anti-HBs level, HBeAg/anti-HBe routine blood test, liver function, renal function will be tested piror to delivery and postpartum 2,6,12 weeks. plasmacytoid dendritic cells(pDCs) and natural killer(NK)cells,CD4＋T cells and regulatory T (Treg) cells were detected by flow cytometry. Plasma cytokines Interferon-alpha 2(IFN-α2) / Interferon-gamma (IFN-γ) / Transforming growth factor beta1 (TGF-β1) / Interleukin-2 (IL-2) / Interleukin-6 (IL-6)/Interleukin-10(IL-10) / Interleukin-17A (IL-17A) / tumor necrosis factor-α1(TNF-α1)were measured by Luminex at the above time point except 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* pregnants who were positivity for serum HBsAg for more than 6 months and HBeAg , HBV DNA >106IU/mL/undetectable HBVDNA ,alanine aminotransferase (ALT) below 35 IU/mL (ULN=40IU/mL) and no received nucleoside analogue antiviral therapy

Exclusion Criteria:

* compensated cirrhosis,hepatic adipose infiltration,ICP. hypertension ,heart disease. postpartum hemorrhage. pregnants who were co-infected with hepatitis A,C,D,E,or HIV;syphilis,Epstein-Barr virus.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: In this trial, pregnants who were positivity for serum HBsAg for more than 6 months and HBeAg , HBV DNA >106IU/mL, alanine aminotransferase (ALT) below 35 IU/mL (ULN=40IU/mL) and no received nucleoside analogue antiviral therapy were enrolled into group A, In addition ,the CHB infection pregnants with undetectable HBVDNA were enrolled into group B(control group).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-01 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
the change of pDCs/ NK/CD4＋T/ Treg cells | in late pregnancy and postpartum 6,12weeks
  the immune function of CHB infecion pregnant women will be evaluated by pDCs/ NK/CD4＋T/ Treg cells
the change of IFN-α2 / IFN-γ)/ TGF-β1 /IL-2 / IL-6/ IL-10 / IL-17A / TNF-α1 | in late pregnancy and postpartum 6,12weeks
  the immune function of CHB infecion pregnant women will be evaluated by IFN-α2 / IFN-γ)/ TGF-β1 /IL-2 / IL-6/ IL-10 / IL-17A / TNF-α1

SECONDARY OUTCOMES:
the change of HBVDNA levels (IU/ML) | in late pregnancy and postpartum 2,6,12weeks
  the prevalence of hepatitis in postpartum pregnant women with chronic hepatitis B virus infection will be evaluated by HBV markers and HBV DNA levels and liver function
the change of ALT levels(U/L) | in late pregnancy and postpartum 2,6,12weeks
  the prevalence of hepatitis in postpartum pregnant women with chronic hepatitis B virus infection will be evaluated by HBV markers and HBV DNA levels and liver function
the change of AST levels(U/L) | in late pregnancy and postpartum 2,6,12weeks
  the prevalence of hepatitis in postpartum pregnant women with chronic hepatitis

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China